CLINICAL TRIAL: NCT03890224
Title: Respiratory Support in Chronic Obstructive Pulmonary Disease (COPD) Patients After Acute Exacerbation With Monitoring the Quality of Support
Brief Title: Respiratory Support in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinact (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Fondation du Souffle (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: R2M; 2018-A01872-53 (Other: ID-RCB)
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD Exacerbation
Keywords: Respiratory Support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Rescue2-monitor is an open-label, prospective randomized, controlled, superiority clinical trial, performed in patients with hypercapnic chronic obstructive pulmonary disease post-acute hypercapnic exacerbation. Four arms (distributed between groups at a ratio of 1:1:1:1) will be compared: no home NIV 'hospital NIV' (control group) versus any of 3 modalities of home NIV (experimental groups). The 3 experimental treatments are Nocturnal home NIV 'non-targeted home NIV', Nocturnal home NIV with high monitoring 'targeted home NIV', and 'rescue home NIV'.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): no home non-invasive ventilation (NIV), only hospital NIV
- Non-targeted home NIV (Active Comparator): Nocturnal home non-invasive ventilation (NIV)
  Interventions: Device: home ventilators
- Targeted home NIV (Active Comparator): Nocturnal home non-invasive ventilation (NIV) with high monitoring
  Interventions: Device: home ventilators
- Rescue home NIV (Active Comparator): home non-invasive ventilation (NIV) on demand
  Interventions: Device: home ventilators

INTERVENTIONS:
Device: home ventilators — The 3 test treatments are home non-targeted NIV, home targeted NIV and rescue home NIV. COPD patients will be equipped with home ventilators and fitted with either nasal, oronasal or facial masks. All the ventilators used will be CE marked.
  Arms: Non-targeted home NIV; Rescue home NIV; Targeted home NIV

SUMMARY:
The hypothesis of this study is that any of 3 modalities of home non- invasive ventilation (NIV) compared to 'no NIV' (=hospital NIV) will reduce re-admission to hospital or death in COPD patients who remain persistently hypercapnic following an exacerbation requiring NIV.

DETAILED DESCRIPTION:
By 2020, chronic obstructive pulmonary disease (COPD) is expected to be the 3rd leading cause of death in the world, especially in countries of middle to high income, like EU. Despite the improvements in survival by using acute non- invasive ventilation (NIV) to treat patients with exacerbations of COPD complicated by acute hypercapnic respiratory failure (AHRF), these patients are at high risk of re-admission and further life-threatening events. Furthermore, in a recent study of 110 patients who had AHRF (RESCUE study, Struik, Thorax 2014), at one year after discharge 65% had another life-threatening event, and 49% had died. New recent data suggests that NIV at home can reduce re-admissions (HMV-LTOT, Murphy, JAMA 2017), but in a small proportion of patients, and with a high level of expertise. There is an urgent need to develop strategies to reduce the number and severity of exacerbations of COPD. With healthcare objectives and budget constraints, telemonitoring of COPD patients is an important challenge in most European countries. RESCUE2-Monitor is the next step. This European trial (currently, France, Spain and Portugal) will test the hypothesis that home NIV, with a highly adapted ventilatory strategy (hereafter referred to as 'TARGETED VENTILATION'), compared to no home NIV (only hospital NIV), to non-targeted home NIV or to rescue home NIV will reduce re-admission to hospital or death in COPD patients, is possible using e-medicine, and will reduce costs of health.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with COPD, GOLD C or D and Forced expiratory volume in one second (FEV1)<65%;
* 2) AHRF (pH<7,35 and PaCO2≥45mm Hg (≥6kPa) treated more than 24h with Ventilation (non-invasive or invasive);
* 3) 48h to 2 weeks with pH>7.35, and PaCO2>45 (>6kPa) after NIV withdrawal, during daytime at rest without oxygen or ventilatory support (or with O2 if patients are not able to avoid O2 with immediate desaturation below 80%).

Exclusion Criteria:

1. Patient treated with chronic NIV or continuous positive airway pressure (CPAP) device, with ongoing treatment;
2. Primary diagnosis of restrictive lung disease causing hypercapnia i.e. obesity hypoventilation and chest wall disease, however these patients will be included if the "FEV1/Forced vital capacity (FVC)" ratio is <60% and the FEV1 <50% if the predominant defect is considered to be obstructive by the center clinician;
3. BMI > 35 kg/m2;
4. Sedative medication causing hypercapnia (> 3 drugs or more than 20mg of morphine/day);
5. Polygraphic diagnosis of Obstructive Sleep Apnoea Syndrome (AHI>30/h (French criteria);
6. Cognitive impairment that would prevent informed consent into the trial
7. Pregnancy;
8. Tobacco use < 10 pack-year;
9. Psychiatric disease necessitating anti-psychotic medication, ongoing treatment for drug or alcohol addiction, persons of no fixed abode post-discharge;
10. Unstable coronary artery syndrome;
11. Age <18 years;
12. Inability to comply with the protocol;
13. Expected survival<12 months due to any situation other than COPD disease;
14. Duration of ICU stay>10 days;
15. No affiliated to national health insurance;
16. Measure of legal protection (guardianship, wardship or judicial protection) for patients over the age of majority.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
admission-free survival | 0-36 months
  defined as time from randomisation to hospital admission in relation with severe exacerbation of COPD or death from any cause, whichever event occurred first, estimated using the Kaplan-Meier method. If neither event occurs, then time will be taken from day randomisation to the last known follow up visit. If withdrawal occurs prior to death, time will be taken from the day of randomisation to day of withdrawal.

SECONDARY OUTCOMES:
Overall survival | 0-36 months
  estimated using the Kaplan-Meier method
Frequency of exacerbations requiring hospitalization | 12 months
  The number of patients that experience one or more exacerbations resulting in hospitalisation
Frequency of exacerbations resulting in physician directed treatment | 12 months
  The number of patients that experience an exacerbation resulting in physician directed treatment, self-management or no treatment change;
Assessment of Exacerbation based on changes in arterial pressure of carbon dioxide | 0, 1, 3, 6, 12, 18, 24, 30 and 36 months
  Change in arterial partial pressure of carbon dioxide (PaCO2) in mmHg
Assessment of Exacerbation based on changes in arterial partial pressure of oxygen | 0, 1, 3, 6, 12, 18, 24, 30 and 36 months
  Change in arterial partial pressure of oxygen (PaO2) severe respiratory insufficiency in mmHg
Assessment of Quality of life with St George's respiratory questionnaire | 0,1, 3, 6, 24 and 36 months
  Evolution of scores obtained at the St George's respiratory questionnaire. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
Assessment of Quality of life with Severe Respiratory Insufficiency Questionnaire | 0,1, 3, 6, 24 and 36 months
  Evolution of scores obtained at the Severe Respiratory Insufficiency Questionnaire The SRI consists of seven subscales covering 49 items: Respiratory Complaints (SRI-RC), Physical Functioning (SRI-PF), Attendant Symptoms and Sleep (SRI-AS), Social Relationships (SRI-SR), Anxiety (SRI-AX), Psychological Well-Being (SRI-WB), and Social Functioning (SRI-SF). These seven subscales can be summarised to one Summary Scale (SRI-SS). All items relate to the patients' circumstances of the last week. Rating for each item is provided by a five-point Likert-scale, a scaling method which measures either positive or negative responses to a given statement with five possible grading steps ranging from "strongly agree" to "strongly disagree". Higher scores are attributed to better Health Related Quality of life.
Assessment of Quality of life with SF-36 | 0,1, 3, 6, 24 and 36 months
  Evolution of scores obtained at SF-36 questionnaire. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Assessment of Quality of life with the 5-level EQ-5D version | 0,1, 3, 6, 24 and 36 months
  Evolution of scores obtained at the EQ5D5L, a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal1
Assessment of Quality of life with the Charlson Comorbidity Index | 0,1, 3, 6, 24 and 36 months
  Evolution of the Charlson Comorbidity Index, a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD). A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
Assessment of Quality of life with the COPD Assessment Test (CAT) | 0,1, 3, 6, 24 and 36 months
  Evolution of the CAT score. The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time.
Assessment of Quality of sleep with Pittsburgh Sleep Quality Index | 0,1, 3, 6, 24 and 36 months
  Evolution of the Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Assessment of Quality of sleep with Epworth Sleepiness Scale | 0,1, 3, 6, 24 and 36 months
  Evolution of the score of Epworth Sleepiness Scale. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought
Assessment of dyspnea with Modified Medical Research Council (mMRC) scale | 0,1, 3, 6, 24 and 36 months
  Evolution of the mMRC score. Dyspnea in daily living was evaluated by the mMRC scale which consists in five statements that describe almost the entire range of dyspnea from none (Grade 0) to almost complete incapacity (Grade 4)
Adverse events (AEs) frequency | 0, 3, 6, 12, 18, 24 and 36 months
  Serious adverse events (SAEs) occurrence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Gonzalez, MD, Principal Investigator — Hôpital Pitié Salpêtrière-Charles Foix, Paris, France ,
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière-Charles Foix, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rescue2-monitor group. Respiratory support in COPD patients after acute exacerbation with monitoring the quality of support (Rescue2-monitor): an open-label, prospective randomized, controlled, superiority clinical trial comparing hospital- versus home-based acute non-invasive ventilation for patients with hypercapnic chronic obstructive pulmonary disease. Trials. 2020 Oct 22;21(1):877. doi: 10.1186/s13063-020-04672-w. PMID 33092618